CLINICAL TRIAL: NCT05574439
Title: Young Adults With Early-onset Obesity Treated With Semaglutide -The RESETTLE Study
Brief Title: Young Adults With Early-onset Obesity Treated With Semaglutide
Acronym: RESETTLE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Signe Torekov (Other)
Collaborators: University of Leeds (Other); Karolinska Institutet (Other); Holbaek Sygehus (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Signe Torekov, Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U1111-1215-8606; 2019-002274-31 (EudraCT Number)
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Obesity, Adolescent
Keywords: GLP-1 RA; Semaglutide; Weight loss; Treatment resistant
MeSH Terms: conditions — Pediatric Obesity; Weight Loss | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Four groups will be identified based on their previous response to structured lifestyle interventions. Non-responders (group A) and insufficient responders (group B) are randomized 2:1 to either Semaglutide 2.4 mg/ week sc or placebo for 68 weeks. Group C (excellent responders) and Group D (population-based reference group with normal weight development) will attend baseline examinations only and not undergo intervention.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The above-mentioned are masked in terms of semaglutide/placebo. Statistical analysis of primary outcome will be blinded to the assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Non-responders: TCOC+ semaglutide (Active Comparator): Semaglutide: 2.4 mg/week SC, concentration: 3.0 mg/ml) in combination with TCOC treatment (i.e. diet/weight consultations).
  Interventions: Behavioral: TCOC treatment; Drug: Semaglutide 3 mg/ml
- Non-responders: TCOC+ placebo (Placebo Comparator): Placebo: 2.4 mg/week SC in combination with TCOC treatment (i.e. diet/weight consultations).
  Interventions: Behavioral: TCOC treatment; Drug: Placebo (Semaglutide 3 mg/ml)
- Insufficient responders: TCOC+ semaglutide (Active Comparator): Semaglutide: 2.4 mg/week SC, concentration: 3.0 mg/ml) in combination with TCOC treatment (i.e. diet/weight consultations).
  Interventions: Behavioral: TCOC treatment; Drug: Semaglutide 3 mg/ml
- Insufficient responders: TCOC+ placebo (Placebo Comparator): Placebo: 2.4mg/week SC in combination with TCOC treatment (i.e. diet/weight consultations).
  Interventions: Behavioral: TCOC treatment; Drug: Placebo (Semaglutide 3 mg/ml)
- Excellent Responders and Population-based reference group (No Intervention): No intervention.

INTERVENTIONS:
Behavioral: TCOC treatment — The TCOC protocol is a chronic care, family-based and multidisciplinary childhood obesity treatment program involving behavior-changing techniques, based on current guidelines for best-practice and authoritative recommendations involving a multidisciplinary tertiary team of health care professionals.
  Arms: Insufficient responders: TCOC+ placebo; Insufficient responders: TCOC+ semaglutide; Non-responders: TCOC+ placebo; Non-responders: TCOC+ semaglutide
Drug: Semaglutide 3 mg/ml — Participants will be instructed to initiate at 0.24 mg SC once weekly for 4 weeks, and in 4 week intervals, increase the dose until a dose of 2.4 mg is reached. In case of prolonged side effects the dose may be adjusted to lower than 2.4mg/week.
  Arms: Insufficient responders: TCOC+ semaglutide; Non-responders: TCOC+ semaglutide
Drug: Placebo (Semaglutide 3 mg/ml) — Participants will be instructed to initiate at 0.24 mg SC once weekly for 4 weeks, and in 4 week intervals, increase the dose until a dose of 2.4 mg is reached. In case of prolonged side effects the dose may be adjusted to lower than 2.4mg/week.
  Arms: Insufficient responders: TCOC+ placebo; Non-responders: TCOC+ placebo

SUMMARY:
Introduction:

The increasing prevalence of obesity is particularly pronounced among adolescents. Currently available treatment options consist of structured lifestyle interventions. However, 25 % of adolescents do not respond to lifestyle treatment, why new effective treatment strategies are needed. Therefore, the aim of this study is to investigate the effect of lifestyle interventions combined with the GLP-1 receptor agonist semaglutide to young adults with otherwise treatment resistant obesity.

Methods and analysis:

This is an investigator-initiated, randomized, placebo-controlled trial. 180-270 young adults (age 18-28) will be recruited from The Childrens Obesity Clinic (TCOC), Department of Pediatrics, Holbæk Hospital. Based on their previous response to the TCOC protocol the participants will be divided in four groups:

Group A: Non-responders: 55-85 young adults with obesity (BMI≥30 kg/m2) who have not reduced adiposity, defined as BMI SDS reduction <0.1, during the structured lifestyle counselling as children.

Group B: Insufficient responders: 55-85 young adults who have reduced adiposity, defined as BMI SDS reduction >0.25, during the structured lifestyle counselling as children but still have obesity as young adults (BMI≥30 kg/m2)

Group C: Excellent responders: 35-50 young adults, who have reduced adiposity, defined as BMI SDS reduction >0.5, during the structured lifestyle counselling as children and no longer have obesity as young adults (BMI<30 kg/m2)

Group D: Population-based reference group (normal weight development): 35-50 young adults, who have participated in The Holbaek Study as children.

Group A and B are randomized 2:1 to either semaglutide or placebo for 68 weeks. Group C and D will attend baseline examinations only and not undergo intervention. The primary endpoint is change in BMI from randomization to end-of-treatment.

Ethics and dissemination: The trial has been approved by the Danish Medicines Agency (EudraCT 2019-002274-31) and by the ethical committee of the Capital Region of Denmark (H-20039422). The trial will be conducted in agreement with the Declaration of Helsinki and monitored to follow the guidelines for good clinical practice. Results will be submitted for publication in international peer-reviewed scientific journals.

DETAILED DESCRIPTION:
Background:

The prevalence of obesity in adolescents has increased markedly in the past decades, thus entailing increased cumulative incidences of type 2 diabetes, cardiovascular disease, and chronic kidney disease (1). Adolescents with obesity are at a substantially elevated risk of developing morbid obesity and type 2 diabetes in early adulthood (2,3) and a recent large scale meta-analysis revealed that mortality increased approximately log-linearly with BMI over 25.0 kg/m² in all continents; and that this increment was greater in younger than older people (4). Furthermore, obesity increase the risk of stigmatization with respect to social relationships, entry into the job market, reduced self-esteem and other psychological problems (5). Thus, adolescents with obesity require particular medical attention.

Since 2008, The Childrens Obesity Clinic (TCOC), Department of Pediatrics, Copenhagen University Hospital Holbæk has treated more than 4000 children and adolescents with overweight or obesity using the TCOC protocol which includes regular counselling on diet, exercise, lifestyle and general health. The TCOC protocol has proven successful with a reduction in BMI standard deviation score (SDS) after 1.5 years of treatment obtained in 74% of the children and adolescents (6). In addition, significant improvements in lipid profile (7) the degree of hypertension (8), hepatic steatosis (9) and the presence of visceral fat (9) have been reported.

However, approximately one in four of the children following the TCOC protocol do not achieve a reduction in BMI SDS. Furthermore, for the majority of children who reduce BMI SDS, obesity remains and represents a medical and personal issue. Lifestyle intervention is the method of choice for children with obesity, however, new effective treatment strategies for non-responders are urgently required.

Glucagon-like peptide-1 (GLP-1) is secreted from endocrine cells in the intestine upon meal intake and reduces blood glucose and food intake in a dose-dependent manner (10-13). It has previously been shown that 1) people with obesity have impaired GLP-1 secretion already in the overweight state, indicating that low concentrations of GLP-1 may be part of obesity development (14), 2) weight loss induces a marked increase in GLP-1 response and this increase is part of a successfully maintained weight loss of >10 kg (15), 3) treatment with a GLP-1 receptor agonist (GLP-1 RA) facilitates long term weight loss maintenance (13 kg) accompanied by substantial improvement in metabolic health, compared to similar diet-induced weight loss maintenance (15-17),4) appetite sensation and eating behavior are important factors in maintenance of weight loss (18,19). Pathogenic mutations in the appetite-regulating melanocortin-4 receptor represent the most common cause of early-onset monogenic obesity that has been shown to be a type of obesity that is more resistant to lifestyle interventions (20) and even to bariatric surgery (21). Interestingly, this population is responsive to treatment with GLP-1 RA (liraglutide 3.0 mg daily) (22). This indicates that GLP-1 RAs can overrule lifestyle modification-resistant obesity due to the appetite-inhibiting effect. A new GLP1-1 RA (semaglutide) was approved by the European Medical Agency (EMA) for weight management in adults with obesity in January 2022. Placebo subtracted weight loss with semaglutide 2.4 mg was 13.9 % compared to 4.5% with liraglutide 3.0 mg after 68 weeks in adults with overweight or obesity (23). Thus, semaglutide has a potentially larger treatment effect also in young adults with childhood onset obesity. The treatment effect of semaglutide 2.4 mg in young adults with lifestyle-treatment-resistant childhood onset obesity is currently unknown, why the outcomes of this study is of high clinical and socioeconomic relevance.

Study hypothesis:

Treatment with a GLP-1 RA will facilitate weight loss in young adults with and without treatment-resistant childhood-onset obesity.

Objectives:

A) To treat young adults with obesity, who have been resistant to structured lifestyle intervention (TCOC protocol), with the GLP-1 RA, semaglutide 2.4 mg/ week.

B) To treat young adults with obesity, who have responded insufficiently to the structured lifestyle intervention (TCOC protocol) and still have obesity, with semaglutide 2.4 mg/ week.

C) To identify underlying mechanisms of lifestyle-untreatable versus treatable childhood-onset obesity.

D) Assess the efficacy of an exercise-based strategy to discontinue obesity medication while sustaining a healthy body composition in youth with childhood-onset obesity.

Endpoints:

Primary endpoint:

1. Change in BMI (weight in kg/height in m^2) from before to after semaglutide treatment compared to placebo.

Secondary endpoints (changes from before to after semaglutide treatment compared to placebo):

1. Body composition (fat mass, fat percentage, fat-free mass, visceral fat, liver fat)
2. Changes in metabolic health:

   (e.g. glucose and insulin for HOMA-IR and Matsuda index, HbA1c, lipids i.e. cholesterol, HDL, LDL, triglycerides, FFA glucose-tolerance status, blood pressure, pulse, and hip and waist circumference, and calculate metabolic syndrome prevalence and metabolic syndrome z-score, and waist-to-height ratio.
3. Body weight
4. Proportion with a reduction in body weight of at least 5%, 10%, 15%, and 20%

The changes in endpoints from baseline (randomization) to after 68 weeks of treatment will be analyzed for all participants treated with semaglutide compared with all participants receiving placebo, and separately in non-responders and insufficient responders to the TCOC protocol, semaglutide compared with placebo.

Other prespecified endpoints:

To determine the effect of GLP-1 RA treatment, and compare data between the two intervention groups, excellent responders and a population-based reference group with normal weight development for the above-mentioned and following outcomes:

1. Questionnaires will be given to the participants to determine self-rated quality of life (SF-36 and PedsQL), eating habits (three-factor eating questionnaire, BED-Q), physical activity (IPAQ), food preferences, self-efficacy (G-SES), sleep quality (PSQI), and appetite (VAS)
2. Conventional Magnetic resonance imaging (MRI) and spectroscopy is used to assess effects on fat deposits in liver, viscera, and muscle. Site-specific bone-measurements, collection of bone markers (CTX and P1NP), and DEXA scans will be performed to assess bone-health.

2. To explore the effects on appetite regulation and systemic markers of immuno-metabolism: Hormonal appetite regulation will be measured during meal tests and fasting (eg. GLP-1, Peptide YY, Glucagon, Leptin, Ghrelin, Liver-Expressed Antimicrobial Peptide 2 (LEAP2), Adiponectin, GDF-15, N-lactoyl-phenylalanine, neurotensin, neprilysin) using our standard methodologies. In plasma samples various biomarkers of inflammation will be measured (e.g., sCD163, hsCRP, IL1, IL2, IL4, IL8, IL10, IL12p70, IL13, IL-1Rap IL-6, TNF-α, SAA1, SAA2, ORM1, ORM2, ICAM-1, VCAM-1, tPA, vWF) and oxidation (eg malonyldialdehyde, F2-Isoprostanes, etc.), IPS, sphingolipids, and metabolomics using plasma metabolomics and proteomics technique. We will also measure metabolic disruptors (e.g., per- and polyfluorinated substances (PFAS)) and store cells for induction of pluripotent stem cell cultures (iPSC), and perform peripheral blood mononuclear cells (PBMNCs) isolation, including DNA collection.

3. To explore the effects on immuno-metabolic profile in human subcutaneous (sc) adipose tissue and gene expression profile of adipose tissue and in circulating inflammatory cells (PBMNCs),we will perform RNA sequencing (Illumina sequencing 30 million paired-end reads/sample) and determine the changes in pro-inflammatory (e.g. IL-6, IL1b, MCP-1, resistin, leptin, chemerin, etc.) and anti-inflammatory (e.g. adiponectin) adipocytokines, and in adipocyte differentiation markers such as FAB4, CABPA and PPAR-γ as well as markers of macrophages infiltration (CD163, CD68) and M1/M2 phenotype of them such as CD40, CCR7, CD207 etc. (all by qRTPCR).

4. To explore the effect on food preferences and appetite sensation: Food preferences are assessed by a picture display test where standardized pictures of food items are shown. Subjective appetite sensations will be obtained during a fixed standardized meal using electronic visual analogue scales (VAS) to record hunger, satiety, fullness, prospective food consumption, desire to eat something fatty, salty, sweet or savory, and palatability of the meals.

5. To explore the effect on brain structure and activity using magnetic resonance imaging (MRI): Brain MRI will be conducted in a subset of participants by trained personnel at the Neurobiological Research Unit, at Copenhagen University Hospital, Rigshospitalet. Pre- and post-meal scans will be performed. From brain MRI we will examine functional connectivity (whole-brain, seed-to-voxel analysis (with the hypothalamus as the primary seed and additional regions of interest (ROI)), and ROI-to-ROI analysis), resting-state networks, brain age, and structural measures such as gray matter volume. Resting-state networks will be examined using Independent Component Analysis in the CONN toolbox. Structural measures, including gray matter volume, will be obtained with FreeSurfer software, and brain age will be estimated using the Pyment software package. Each brain MRI session will last approximately one hour.

6. To explore the genetic risk scores correlated to treatment response: All participants are chip genotyped to define polygenic risk scores. DNA material will be extracted from blood samples. The Infinium Global Screening Array will be used to analyze the array with Illumina Genome Studio before the bioinformatic removal of SNPs containing genes mentioned in the "American College Medical Genetics and Genomics" List.

7. To explore the effect on the microbiota: The microbiome will be measured in fecal and saliva samples of participants. Furthermore, fecal and saliva samples were collected from the same individuals when they were children with obesity, allowing for comparison of potential differences already evident in childhood that may indicate later treatment response to lifestyle change and GLP-1RA treatment.

8. To explore the effect on metabolomics in urine: Urine samples are collected at the two test days and will be stored frozen for later analyses for potential changes in the metabolomic profile.

9. Psycho-social aspects of obesity development and treatment response We will evaluate the effect of adversity measures across upbringing and current living conditions and explore eating practices and individual weight trajectories in relation to psychological and social factors.

10. A physical activity tracker will be worn on the wrist throughout the study period to assess habitual physical activity and sleep habits.

11. To explore the effect of post medication phase on limiting weight and fat regain: We will investigate whether a post medication program after GLP-1RA discontinuation, comprising data-driven supervised exercise, sleep, and healthy eating behaviour, can limit weight and fat regain and limit deterioration of metabolic health. We will perform DEXA scans 26 weeks after medication termination to investigate changes in body fat percentage, fat mass, and lean mass. We will investigate changes in the outcomes mentioned above and grip strength.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-28 years
* The period from the initial treatment with TCOC protocol until inclusion in the study must be within 15 years.
* Group A: BMI≥30. Non-responders: No BMI SDS reduction (≤0.1 BMI SDS) during TCOC protocol for more than one year and still have obesity.
* Group B: BMI≥30. Insufficient responders: BMI SDS reduction ≥0.25 BMI SDS during TCOC protocol for more than one year, but still have obesity.
* Group C: BMI≤30. Excellent responders: BMI SDS reduction ≥0.5 BMI SDS during TCOC protocol for more than one year and no longer have obesity.
* Group D: Young adults who have participated in The Holbaek Study and have had normal weight development during childhood

Exclusion Criteria:

* Participants diagnosed with known serious chronic illness including type 1 or 2 diabetes (or a randomly measured fasting plasma glucose >7 mmol/l)
* Angina pectoris, coronary heart disease, congestive heart failure (NYHA III-IV)
* Severe renal impairment (creatinine clearance (GFR) <30 mL/min)
* Severe hepatic impairment
* Inflammatory bowel disease
* Diabetic gastroparesis
* Cancer
* Chronic obstructive lung disease
* Severe psychiatric disease, a history of major depressive or other severe psychiatric disorders
* Use of medications causing clinically significant weight gain or loss
* Previous bariatric surgery
* A history of idiopathic acute pancreatitis
* A family or personal history of multiple endocrine neoplasia type 2 or familial medullary thyroid carcinoma
* Pregnancy, expecting pregnancy or breastfeeding. If a study participant is in doubt whether she could be pregnant, a urine pregnancy test is performed. Women with reproductive potential who are not using adequate contraceptive methods (combined oral contraceptive pill, progestin-only contraceptive pill, condoms, intrauterine device, injection, implant, or sterilization). Adequate contraception must be used throughout the study period and at least 2 months after discontinuation of trial medication (semaglutide will be present in the circulation for 5-7 weeks after the last dose).
* Allergy to any of the ingredients/excipients of the study medication: Semaglutide, disodium phosphate dihydrate, propylene glycol, phenol, hydrochloric acid, sodium hydroxide.
* Exclusion criteria for MRI: Pacemaker, claustrophobia, metal splinters or any other magnetic devices that cannot be removed prior to the scan (Participants can join the trial without MR scan)

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in BMI (weight in kg/height in m^2) | Change from baseline to end-of-treatment (68 weeks)
  Weight will be measured to the nearest 0.1 kg. The same set of scales should ideally be used throughout the trial. Weight should be measured in a fasting state without shoes and wearing light indoor clothes. Height will be measured to the nearest 0.1 cm.

SECONDARY OUTCOMES:
Change in body composition (fat mass) | Change from baseline to end-of-treatment (68 weeks)
  Dual-energy X-ray absorptiometry scans will be performed in fasting state to measure body fat mass (kg).
Change in body composition (fat percentage) | Change from baseline to end-of-treatment (68 weeks)
  Dual-energy X-ray absorptiometry scans will be performed in fasting state to measure body fat percentage (%).
Change in body composition (fat free mass) | Change from baseline to end-of-treatment (68 weeks)
  Dual-energy X-ray absorptiometry scans will be performed in fasting state to measure fat-free mass (kg).
Change in visceral fat and liver fat | Change from baseline to end-of-treatment (68 weeks)
  MRI will be performed in fasting state to measure fat content
Change in metabolic syndrome | Change from baseline to end-of-treatment (68 weeks)
  z-score
Change in waist-to-height ratio | Change from baseline to end-of-treatment (68 weeks)
  waist-to-height ratio
Compare BMI (weight in kg/height in m^2), body composition, body weight, and metabolic health between population-based reference group, excellent responders, non-responders and insufficient responders. | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  Dual-energy X-ray absorptiometry scans will be performed in fasting state to measure fat mass and lean mass (kg)
Change in body weight | Change from baseline to end-of-treatment (68 weeks)
  Body weight change and proportion with at least 5%, 10%, 15%, and 20%
Change in metabolic syndrome | Change from baseline to end-of-treatment (68 weeks)
  Prevalence (%)

OTHER OUTCOMES:
HOMA-IR | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  Fasting insulin (μU/mL) * fasting glucose (mmol/L) / 22.5
Matsuda Index | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  10000/sqrt(fasting glucose * fasting insulin * mean glucose * mean insulin)
Plasma Glucose | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  mmol/L
Plasma Insulin | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  pmol/L
HbA1c | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  mmol/mol
Lipids | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  Cholesterol (Total, HDL, LDL, VLDL) and triglycerides (TG)) (mmol/L)
Free Fatty Acids | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  umol/L
Waist and hip circumference | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  Waist circumference, the midpoint between lowest rib and iliac crest, and hip circumference, the level of the great trochanters, will be measured in duplicate to the nearest 0.1 cm after gentle expiration.
Blood pressure | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  Blood pressure (systolic/diastolic) will be measured in duplicate from the non-dominant arm with a digital blood pressure monitor in sitting position after at least 5 min of rest (mmHg).
Heart rate | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  Heart rate (bpm)
Ectopic fat accumulation in liver, viscera and muscle | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  Magnetic resonance imaging (MRI) and spectroscopy
Brain structure and function | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  Magnetic resonance imaging (MRI) will be performed in the fasting and fed states to assess brain structure and function.
Bone mineral density | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  Dual energy x-ray absorptiometry (DEXA) (g/cm^2)
Bone markers | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  CTX (ng/l) and P1NP (µg/L)
Hormonal appetite regulation during meal tests and in fasting | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  GLP-1, Peptide YY, Glucagon, Leptin, Ghrelin, LEAP2, Adiponectin, GDF-15, N-lactoyl-phenylalanine, neurotensin, neprilysin
Systemic biomarkers of inflammation | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  e.g. sCD163, hsCRP, IL1, IL2, IL4, IL8, IL10, IL12p70, IL13, IL-1Rap IL-6, TNF-α, SAA1, SAA2, ORM1, ORM2, ICAM-1, VCAM-1, tPA, vWF) and oxidation (e.g., malonyldialdehyde, F2-Isoprostanes, etc.), IPS, sphingolipids, metabolomics using plasma metabolomics, and proteomics
Systemic biomarkers of oxidation | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  Malonyldialdehyde and F2-Isoprostanes
Immunometabolic profile of subcutaneous adipose tissue | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  Pro-inflammatory (e.g. IL-6, IL1b, MCP-1, resistin, leptin, chemerin, etc.) and anti-inflammatory (e.g. adiponectin) adipocytokines.
RNA sequencing on subcutaneous adipose tissue | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  Illumina sequencing
Food preferences | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  Leeds Food Preference Questionnaire (LFPQ)
Subjective appetite sensation | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  Electronic visual analogue scales (VAS) (0-100 scale)
Genetic risk score correlated to treatment response | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  From blood samples, DNA material will be extracted and analyzed using the Infinium Global Screening Array and Illumina Genome Studio
Gut microbiota composition | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  Collection of saliva and fecal samples and extraction of genomic DNA
Metabolomics in urine | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  Urine samples
Metabolomics in plasma | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  Metabolomics technique
Proteomics in plasma | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  Proteomics technique
Health-related quality of life | Change from baseline to end-of-treatment (68 weeks)
  SF-36 component scores
Psycho-social aspects of obesity development and treatment response by qualitative content analysis of semi-structured interviews | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  Open-ended semi-structured interviews will be conducted to measure adversity, resources, eating practices, and individual weight trajectories (score)
Eating behavior | Baseline comparison and change from baseline to end-of-treatment (68 weeks)
  Three-factor eating questionnaire (0-100 scale where higher score means a better outcome)
Systemic levels of metabolic disruptors | Change from baseline to end-of-treatment (68 weeks)
  Measurement of plasma/serum concentrations of metabolic disruptors (e.g. per- and polyfluorinated substances (PFAS))
Induction of pluripotent stem cell cultures (iPSC) | Baseline comparison
  One blood sample from each participant is used for induction of pluripotent stem cell culture (iPSC).
Muscle Strength | Change from 68 weeks to week 94
  Hand grip strength
Physical activity level | Baseline comparison and changes from baseline to end-of-treatment (week 68)
  Measured by wrist-worn activity tracker (min/week)
Sleep | Baseline comparison and changes from baseline to end-of-treatment (week 68)
  Measured by wrist-worn activity tracker (min/night)
Change in body composition after medication (fat percentage) | Week 68 to 94
  Dual-energy X-ray absorptiometry scans will be performed in fasting state to measure body fat percentage (%).
Change in body composition after medication (fat mass) | Week 68 to 94
  Dual-energy X-ray absorptiometry scans will be performed in fasting state to measure body fat mass (kg).
Change in body composition after medication (fat-free mass) | Week 68 to 94
  Dual-energy X-ray absorptiometry scans will be performed in fasting state to measure fat-free mass (kg).
Change in body weight after medication | Change from week 68 to 94
  Body weight change (kg)
Change in waist-to-height ratio after medication | Change from week 68 to 94
  Waist-to-height ratio
Change in visceral fat and liver fat after medication | Change from week 68 to 94
  MRI will be performed in fasting state to measure fat content
Change in metabolic syndrome after medication | Change from week 68 to 94
  z-score
Health-related quality of life after medication | Change from week 68 to 94
  SF-36 component scores (0-100 scale where higher score means a better outcome)
Physical activity level | Baseline comparison and changes from baseline to end-of-treatment (week 68)
  Measured by International Physical Activity Questionnaire (min/week)
Sleep quality | Baseline comparison and changes from baseline to end-of-treatment (week 68)
  PSQI score

CONTACTS AND LOCATIONS:
Overall Officials: Signe S Torekov, Prof, PhD, Study Director — University of Copenhagen; Jens-Christian Holm, Ass. Prof, PhD, Study Chair — Holbæk University Hospital
Locations (2):
- Denmark (2):
  - Holbæk University Hospital, Holbæk, Region Zeeland
  - University of Copenhagen, Department of Biomedical Sciences, Copenhagen

REFERENCES:
- [Background] GBD 2015 Obesity Collaborators; Afshin A, Forouzanfar MH, Reitsma MB, Sur P, Estep K, Lee A, Marczak L, Mokdad AH, Moradi-Lakeh M, Naghavi M, Salama JS, Vos T, Abate KH, Abbafati C, Ahmed MB, Al-Aly Z, Alkerwi A, Al-Raddadi R, Amare AT, Amberbir A, Amegah AK, Amini E, Amrock SM, Anjana RM, Arnlov J, Asayesh H, Banerjee A, Barac A, Baye E, Bennett DA, Beyene AS, Biadgilign S, Biryukov S, Bjertness E, Boneya DJ, Campos-Nonato I, Carrero JJ, Cecilio P, Cercy K, Ciobanu LG, Cornaby L, Damtew SA, Dandona L, Dandona R, Dharmaratne SD, Duncan BB, Eshrati B, Esteghamati A, Feigin VL, Fernandes JC, Furst T, Gebrehiwot TT, Gold A, Gona PN, Goto A, Habtewold TD, Hadush KT, Hafezi-Nejad N, Hay SI, Horino M, Islami F, Kamal R, Kasaeian A, Katikireddi SV, Kengne AP, Kesavachandran CN, Khader YS, Khang YH, Khubchandani J, Kim D, Kim YJ, Kinfu Y, Kosen S, Ku T, Defo BK, Kumar GA, Larson HJ, Leinsalu M, Liang X, Lim SS, Liu P, Lopez AD, Lozano R, Majeed A, Malekzadeh R, Malta DC, Mazidi M, McAlinden C, McGarvey ST, Mengistu DT, Mensah GA, Mensink GBM, Mezgebe HB, Mirrakhimov EM, Mueller UO, Noubiap JJ, Obermeyer CM, Ogbo FA, Owolabi MO, Patton GC, Pourmalek F, Qorbani M, Rafay A, Rai RK, Ranabhat CL, Reinig N, Safiri S, Salomon JA, Sanabria JR, Santos IS, Sartorius B, Sawhney M, Schmidhuber J, Schutte AE, Schmidt MI, Sepanlou SG, Shamsizadeh M, Sheikhbahaei S, Shin MJ, Shiri R, Shiue I, Roba HS, Silva DAS, Silverberg JI, Singh JA, Stranges S, Swaminathan S, Tabares-Seisdedos R, Tadese F, Tedla BA, Tegegne BS, Terkawi AS, Thakur JS, Tonelli M, Topor-Madry R, Tyrovolas S, Ukwaja KN, Uthman OA, Vaezghasemi M, Vasankari T, Vlassov VV, Vollset SE, Weiderpass E, Werdecker A, Wesana J, Westerman R, Yano Y, Yonemoto N, Yonga G, Zaidi Z, Zenebe ZM, Zipkin B, Murray CJL. Health Effects of Overweight and Obesity in 195 Countries over 25 Years. N Engl J Med. 2017 Jul 6;377(1):13-27. doi: 10.1056/NEJMoa1614362. Epub 2017 Jun 12. PMID 28604169
- [Background] Bjerregaard LG, Jensen BW, Angquist L, Osler M, Sorensen TIA, Baker JL. Change in Overweight from Childhood to Early Adulthood and Risk of Type 2 Diabetes. N Engl J Med. 2018 Apr 5;378(14):1302-1312. doi: 10.1056/NEJMoa1713231. PMID 29617589
- [Background] The NS, Suchindran C, North KE, Popkin BM, Gordon-Larsen P. Association of adolescent obesity with risk of severe obesity in adulthood. JAMA. 2010 Nov 10;304(18):2042-7. doi: 10.1001/jama.2010.1635. PMID 21063014
- [Background] Global BMI Mortality Collaboration, Di Angelantonio E, Bhupathiraju ShN, Wormser D, Gao P, Kaptoge S, Berrington de Gonzalez A, Cairns BJ, Huxley R, Jackson ChL, Joshy G, Lewington S, Manson JE, Murphy N, Patel AV, Samet JM, Woodward M, Zheng W, Zhou M, Bansal N, Barricarte A, Carter B, Cerhan JR, Smith GD, Fang X, Franco OH, Green J, Halsey J, Hildebrand JS, Jung KJ, Korda RJ, McLerran DF, Moore SC, O'Keeffe LM, Paige E, Ramond A, Reeves GK, Rolland B, Sacerdote C, Sattar N, Sofianopoulou E, Stevens J, Thun M, Ueshima H, Yang L, Yun YD, Willeit P, Banks E, Beral V, Chen Zh, Gapstur SM, Gunter MJ, Hartge P, Jee SH, Lam TH, Peto R, Potter JD, Willett WC, Thompson SG, Danesh J, Hu FB. Body-mass index and all-cause mortality: individual-participant-data meta-analysis of 239 prospective studies in four continents. Lancet. 2016 Aug 20;388(10046):776-86. doi: 10.1016/S0140-6736(16)30175-1. Epub 2016 Jul 13. PMID 27423262
- [Background] Hebebrand J, Holm JC, Woodward E, Baker JL, Blaak E, Durrer Schutz D, Farpour-Lambert NJ, Fruhbeck G, Halford JGC, Lissner L, Micic D, Mullerova D, Roman G, Schindler K, Toplak H, Visscher TLS, Yumuk V. A Proposal of the European Association for the Study of Obesity to Improve the ICD-11 Diagnostic Criteria for Obesity Based on the Three Dimensions Etiology, Degree of Adiposity and Health Risk. Obes Facts. 2017;10(4):284-307. doi: 10.1159/000479208. Epub 2017 Jul 22. PMID 28738325
- [Background] Mollerup PM, Gamborg M, Trier C, Bojsoe C, Nielsen TR, Baker JL, Holm JC. A hospital-based child and adolescent overweight and obesity treatment protocol transferred into a community healthcare setting. PLoS One. 2017 Mar 6;12(3):e0173033. doi: 10.1371/journal.pone.0173033. eCollection 2017. PMID 28264043
- [Background] Nielsen TR, Gamborg M, Fonvig CE, Kloppenborg J, Hvidt KN, Ibsen H, Holm JC. Changes in lipidemia during chronic care treatment of childhood obesity. Child Obes. 2012 Dec;8(6):533-41. doi: 10.1089/chi.2011.0098. PMID 23181919
- [Background] Hvidt KN, Olsen MH, Ibsen H, Holm JC. Effect of changes in BMI and waist circumference on ambulatory blood pressure in obese children and adolescents. J Hypertens. 2014 Jul;32(7):1470-7; discussion 1477. doi: 10.1097/HJH.0000000000000188. PMID 24733029
- [Background] Fonvig CE, Chabanova E, Ohrt JD, Nielsen LA, Pedersen O, Hansen T, Thomsen HS, Holm JC. Multidisciplinary care of obese children and adolescents for one year reduces ectopic fat content in liver and skeletal muscle. BMC Pediatr. 2015 Dec 30;15:196. doi: 10.1186/s12887-015-0513-6. PMID 26714769
- [Background] Torekov SS, Holst JJ, Ehlers MR. Dose response of continuous subcutaneous infusion of recombinant glucagon-like peptide-1 in combination with metformin and sulphonylurea over 12 weeks in patients with type 2 diabetes mellitus. Diabetes Obes Metab. 2014 May;16(5):451-6. doi: 10.1111/dom.12240. Epub 2013 Dec 10. PMID 24251641
- [Background] Torekov SS, Kipnes MS, Harley RE, Holst JJ, Ehlers MR. Dose response of subcutaneous GLP-1 infusion in patients with type 2 diabetes. Diabetes Obes Metab. 2011 Jul;13(7):639-43. doi: 10.1111/j.1463-1326.2011.01388.x. PMID 21362122
- [Background] Torekov SS, Madsbad S, Holst JJ. Obesity - an indication for GLP-1 treatment? Obesity pathophysiology and GLP-1 treatment potential. Obes Rev. 2011 Aug;12(8):593-601. doi: 10.1111/j.1467-789X.2011.00860.x. Epub 2011 Mar 15. PMID 21401851
- [Background] Flint A, Raben A, Astrup A, Holst JJ. Glucagon-like peptide 1 promotes satiety and suppresses energy intake in humans. J Clin Invest. 1998 Feb 1;101(3):515-20. doi: 10.1172/JCI990. PMID 9449682
- [Background] Faerch K, Torekov SS, Vistisen D, Johansen NB, Witte DR, Jonsson A, Pedersen O, Hansen T, Lauritzen T, Sandbaek A, Holst JJ, Jorgensen ME. GLP-1 Response to Oral Glucose Is Reduced in Prediabetes, Screen-Detected Type 2 Diabetes, and Obesity and Influenced by Sex: The ADDITION-PRO Study. Diabetes. 2015 Jul;64(7):2513-25. doi: 10.2337/db14-1751. Epub 2015 Feb 12. PMID 25677912
- [Background] Iepsen EW, Lundgren J, Holst JJ, Madsbad S, Torekov SS. Successful weight loss maintenance includes long-term increased meal responses of GLP-1 and PYY3-36. Eur J Endocrinol. 2016 Jun;174(6):775-84. doi: 10.1530/EJE-15-1116. Epub 2016 Mar 14. PMID 26976129
- [Background] Iepsen EW, Lundgren J, Dirksen C, Jensen JE, Pedersen O, Hansen T, Madsbad S, Holst JJ, Torekov SS. Treatment with a GLP-1 receptor agonist diminishes the decrease in free plasma leptin during maintenance of weight loss. Int J Obes (Lond). 2015 May;39(5):834-41. doi: 10.1038/ijo.2014.177. Epub 2014 Oct 7. PMID 25287751
- [Background] Lundgren JR, Janus C, Jensen SBK, Juhl CR, Olsen LM, Christensen RM, Svane MS, Bandholm T, Bojsen-Moller KN, Blond MB, Jensen JB, Stallknecht BM, Holst JJ, Madsbad S, Torekov SS. Healthy Weight Loss Maintenance with Exercise, Liraglutide, or Both Combined. N Engl J Med. 2021 May 6;384(18):1719-1730. doi: 10.1056/NEJMoa2028198. PMID 33951361
- [Background] Christensen BJ, Iepsen EW, Lundgren J, Holm L, Madsbad S, Holst JJ, Torekov SS. Instrumentalization of Eating Improves Weight Loss Maintenance in Obesity. Obes Facts. 2017;10(6):633-647. doi: 10.1159/000481138. Epub 2017 Dec 6. PMID 29207396
- [Background] Jensen SBK, Janus C, Lundgren JR, Juhl CR, Sandsdal RM, Olsen LM, Andresen A, Borg SA, Jacobsen IC, Finlayson G, Stallknecht BM, Holst JJ, Madsbad S, Torekov SS. Exploratory analysis of eating- and physical activity-related outcomes from a randomized controlled trial for weight loss maintenance with exercise and liraglutide single or combination treatment. Nat Commun. 2022 Aug 15;13(1):4770. doi: 10.1038/s41467-022-32307-y. PMID 35970829
- [Background] Trier C, Hollensted M, Schnurr TM, Lund MAV, Nielsen TRH, Rui G, Andersson EA, Svendstrup M, Bille DS, Gjesing AP, Fonvig CE, Frithioff-Bojsoe C, Balslev-Harder M, Quan S, Gamborg M, Pedersen O, Angquist L, Holm JC, Hansen T. Obesity treatment effect in Danish children and adolescents carrying Melanocortin-4 Receptor mutations. Int J Obes (Lond). 2021 Jan;45(1):66-76. doi: 10.1038/s41366-020-00673-6. Epub 2020 Sep 13. PMID 32921795
- [Background] Bonnefond A, Keller R, Meyre D, Stutzmann F, Thuillier D, Stefanov DG, Froguel P, Horber FF, Kral JG. Eating Behavior, Low-Frequency Functional Mutations in the Melanocortin-4 Receptor (MC4R) Gene, and Outcomes of Bariatric Operations: A 6-Year Prospective Study. Diabetes Care. 2016 Aug;39(8):1384-92. doi: 10.2337/dc16-0115. Epub 2016 May 23. PMID 27222505
- [Background] Iepsen EW, Zhang J, Thomsen HS, Hansen EL, Hollensted M, Madsbad S, Hansen T, Holst JJ, Holm JC, Torekov SS. Patients with Obesity Caused by Melanocortin-4 Receptor Mutations Can Be Treated with a Glucagon-like Peptide-1 Receptor Agonist. Cell Metab. 2018 Jul 3;28(1):23-32.e3. doi: 10.1016/j.cmet.2018.05.008. Epub 2018 May 31. PMID 29861388
- [Background] Rubino DM, Greenway FL, Khalid U, O'Neil PM, Rosenstock J, Sorrig R, Wadden TA, Wizert A, Garvey WT; STEP 8 Investigators. Effect of Weekly Subcutaneous Semaglutide vs Daily Liraglutide on Body Weight in Adults With Overweight or Obesity Without Diabetes: The STEP 8 Randomized Clinical Trial. JAMA. 2022 Jan 11;327(2):138-150. doi: 10.1001/jama.2021.23619. PMID 35015037

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-10-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT05574439/SAP_001.pdf